CLINICAL TRIAL: NCT05754151
Title: Feasibility and Acceptability of a Mobile Cognitive Behavior Therapy App Targeting Depression and Anxiety in Older Adults
Brief Title: Mobile CBT for Middle Aged and Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Joseph S. Sanchez Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-01025548
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Anxiety Disorders and Symptoms; Depressive Symptoms; Depression
Keywords: Anxiety; CBT; Mobile Application; Cognitive Behavioral Therapy; Depression; Older Adults; Adults
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Masking Description: All participants will receive the same intervention. Therefore, no masking is required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAYA Mobile App (Experimental): Participants receive treatment with the MAYA application for 6 weeks
  Interventions: Behavioral: MAYA Mobile Application

INTERVENTIONS:
Behavioral: MAYA Mobile Application — The mobile cognitive behavioral therapy (CBT) application, MAYA, teaches cognitive behavioral therapy (CBT) techniques including emotion monitoring, cognitive restructuring, mindfulness, exposure and psychoeducation (i.e. information about anxiety and depression). The application includes an interactive dashboard to provide the user with statistics for tracking progress toward their goals. Although the MAYA application is new, its content and structure are similar to how CBT- a well-established and widely used psychosocial intervention - is commonly delivered in the more traditional setting of a psychotherapist's office.

SUMMARY:
This study aims to assess a mobile iPhone app called MAYA for use in middle-aged and older adults with anxiety or mood disorders. The MAYA app is designed to teach coping skills for anxiety and depression that are drawn from cognitive behavioral therapy. Participants will be asked to use the app for at least two days a week, 20 minutes on each day, for six weeks. Participants will have weekly check-ins as well as longer assessments at the beginning of the study, week 3, week 6 (end of treatment), and week 12 (follow up). During assessments, participants will answer brief questionnaires designed to assess their symptoms and impressions of the app. The main hypotheses of the study are that participants will complete most of the assigned sessions and that they will rate their impressions of the app highly. The secondary hypotheses are that symptoms of depression and anxiety will decrease with use of the MAYA app.

DETAILED DESCRIPTION:
There is a growing need for accessible, affordable, research-supported treatments designed for older adults. Older adults face challenges that limit their ability to physically access mental health services; thus, mobile app-based interventions may be particularly appealing to individuals in this age range with anxiety or depression who are unable to access more traditional psychotherapy administered in person by a therapist. Mobile technology has been used previously to deliver mental health services for adults with a variety of psychiatric symptoms (Dennis & O'Toole, 2014).

Anxiety frequently co-occurs with depression, with 72% of individuals with anxiety having experienced a history of depression (Moffitt et al., 2007). Current models conceptualize anxiety and depression as a confluence of three broad symptom categories - physiological hyperarousal, low positive affect, and high negative affect (Clark & Watson, 1991) - that are present to different degrees in different individuals.

This study aims to assess the acceptability, feasibility and efficacy of "MAYA", a mobile cognitive behavioral therapy app for anxiety and mood disorders, in middle aged and older adults. This study will collect pilot data over the course of 12 weeks. As this is a pilot study, all participants will use the same version of the app and there will be no control group. Participants will be asked to use the mobile app for at least two days a week, for at least 20 minutes on each day, for 6 weeks. Participants will have weekly check-ins in person or via a HIPAA-compliant virtual meeting platform (e.g., Zoom) to assess intervention adherence and answer brief questionnaires designed to assess feasibility, acceptability, and mood symptoms at baseline, week 3, week 6 (end of treatment), and week 12 (follow up).

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or older
* Primary diagnosis of an anxiety or depressive disorder as determined by a clinical severity rating score of 4 or greater on the Anxiety Disorders Interview Schedule (ADIS).
* Mini Mental Status Exam (MMSE) no more than 1 SD below the mean score for patient's age and education. If the remote version of the MMSE is used (e.g. during an evaluation on Zoom), the remote MMSE score will be converted to a standard MMSE score.
* Access to an Apple iPhone

Exclusion Criteria:

* Lifetime diagnosis of a bipolar or psychotic disorder.
* Currently in cognitive behavior therapy.
* Change in dose of a psychiatric medication in the past 12 weeks.
* Initiation of psychotherapy in the past 12 weeks.
* Intent or plan to attempt suicide.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the MAYA application as measured by mean uMARS scores at Baseline | Week 1 (Baseline)
  The primary measure to assess accessibility of the MAYA app will be the User Version of the Mobile Application Rating Scale (uMARS). The uMARS is a 26-item questionnaire that evaluates the quality of the mobile health applications with six subscales: engagement, functionality, aesthetics, information, app subjective quality, perceived impact. Scores on the scale can range from 21 to 130, where higher scores represent higher quality of mobile health applications by end-users.
Acceptability of the MAYA application as measured by mean uMARS scores at Midpoint | Week 3 (Midpoint)
  The primary measure to assess accessibility of the MAYA app will be the User Version of the Mobile Application Rating Scale (uMARS). The uMARS is a 26-item questionnaire that evaluates the quality of the mobile health applications with six subscales: engagement, functionality, aesthetics, information, app subjective quality, perceived impact. Scores on the scale can range from 21 to 130, where higher scores represent higher quality of mobile health applications by end-users.
Acceptability of the MAYA application as measured by mean uMARS scores at Endpoint | Week 6 (Endpoint)
  The primary measure to assess accessibility of the MAYA app will be the User Version of the Mobile Application Rating Scale (uMARS). The uMARS is a 26-item questionnaire that evaluates the quality of the mobile health applications with six subscales: engagement, functionality, aesthetics, information, app subjective quality, perceived impact. Scores on the scale can range from 21 to 130, where higher scores represent higher quality of mobile health applications by end-users.
Feasibility of the MAYA application as measured by total number of sessions completed in the MAYA application at Endpoint | Week 6 (Endpoint)
  Total number of sessions completed by the end of the administered intervention
Feasibility of the MAYA application as measured by total number of sessions completed in the MAYA application at Follow Up | Week 12 (Follow Up)
  Total number of sessions completed by the end of the administered intervention

SECONDARY OUTCOMES:
Change in anxiety symptoms as measured by the HAM-A | Baseline, Week 6 (Endpoint), and Week 12 (Follow Up)
  The primary symptom measure for anxiety will be the Hamilton Rating Scale for Anxiety (HAM-A). The HAM-A is a 14-item questionnaire measure of the severity of anxiety symptoms. The items measure both psychic anxiety and somatic anxiety. The scores range from 0 to 56, where higher scores indicate a greater severity of symptoms and lower scores indicate mild to no anxiety symptoms.
Change in depressive symptoms as measured by the MADRS | Baseline, Week 6 (Endpoint), and Week 12 (Follow Up)
  Depression will be measured using the Montgomery-Asberg Depression Rating Scale (MADRS). The MADRS is a 10-item questionnaire measuring the severity of depression symptoms. Scores range from 0 to 60, where higher scores indicate higher severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bress, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No